CLINICAL TRIAL: NCT03875703
Title: Biological Collection for Studying Vaccine-induced Immune Responses
Brief Title: Post-Vaccination Biological Collection
Acronym: BioCol-VIR
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: K170603J
Record Dates: First submitted 2019-01-18; First posted 2019-03-15 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Vaccination; Immune Response
Keywords: Biological Collection; Vaccination; Active Immune Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood & serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Vaccination is a powerful weapon in the fight against infectious diseases, which has led to dramatic reduction in mortality and complications from some diseases. In this respect, vaccination is a real worldwide public health challenge (WHO). Thus, vaccine research benefits from an exponential development of knowledge in immunology and biotechnology. In particular, the advent of recent tools ("omics", new cytometric assays) and the description of new categories of immune cells (Tfh, BReg...) have revolutionized the characterization of immune responses, particularly post-vaccination. To study of the immune response following vaccination remains essential in order to define the immunological correlates to vaccine protection. This response also varies according to parameters related to the vaccine (type, adjuvant, dose, regimen…) and to the vaccinated host (genetics, age, morbidity, treatment …). Analyzing with new generation immune assays, new data on immunological responses post-vaccination from a clinical cohort is therefore essential to better define these correlates.

Objective: To develop new vaccines (HIV, emerging infectious diseases) the investigators use a "System vaccinology" method to decipher the mechanisms of immune responses set up against vaccines currently being developed or marketed, specifically in specific populations (patients with primary immune deficiency, sickle cell patients, solid organ transplanted patients, COPD).

Method: Description of the genetic, molecular and cellular mechanisms of the immune response to vaccines recommended for adults, in particular influenza and pneumococcal vaccines, but also other mandatory vaccines (MMR,...) or vaccine for travelers (yellow fever, ...) as part of routine care in different population categories (healthy subjects, HIV+ subjects, COPD patients, …), using qualitative and quantitative immunological assays: transcriptional analysis of the dynamic innate immune response, analysis of the lymphocytes B & T responses (phenotype, repertoire analysis, functional analysis including T reg and TFH populations, antibody response), genetic analysis in the context of primary immune deficiencies) Conclusion: The data generated will allow the best possible analysis of vaccine responses according to vaccines and vaccinated populations, providing important information for the research developed within the department.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Informed and consented
* Need to be vaccinated for routine care

Exclusion Criteria:

* Person under guardianship or safeguards
* Pregnant or breastfeeding woman
* No affiliation to a health insurance scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who receive a vaccination in the department of Immunology and Infectious Diseases of the Henri Mondor University Hospital (Créteil, France).
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2030-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in transcriptional analysis, analysis of the innate immune response after vaccination | Hour 24 after vaccination
  Transcriptomic analysis performed from whole blood samples

SECONDARY OUTCOMES:
B cell immune response | at Day 0, Day 7, Day 14 and Month 1 after vaccination
  (phenotype, analysis of the repertoire B, functional analysis, antibody response, plasmablastic response)
T cell immune response | at Day 0, Day 7, Day 14 and Month 1 after vaccination
  (phenotype, T repertoire analysis, functional analysis, especially of the Treg and TFH populations)
Specific antibody response to the used vaccines at M1 | at Month 1

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia Gregoire, Study Chair — APHP URC
Locations (1):
- Pr Gallien, Créteil, France